CLINICAL TRIAL: NCT05751512
Title: A Randomized, Open-Label, Multicenter, Phase III Study to Evaluate MRG003 vs Cetuximab/Methotrexate as Second/Third Line of Treatment in Patient With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (RM-SCCHN)
Brief Title: A Study to Evaluate MRG003 vs Cetuximab/Methotrexate in in the Treatment of Patients With RM-SCCHN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-010
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: MRG003; Antibody Drug Conjugate (ADC); SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRG003 (Experimental): MRG003 will be administrated via intravenous infusion at 2.3 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG003
- cetuximab/ methotrexate (Active Comparator): cetuximab (400 mg/m2 for the first week and 250 mg/m2 for subsequent weeks, QW) or methotrexate (40 mg/m2, IV, QW)
  Interventions: Drug: Cetuximab injection; Drug: Methotrexate Injection

INTERVENTIONS:
Drug: MRG003 — Administered intravenously
  Arms: MRG003
Drug: Cetuximab injection — Administered intravenously
  Arms: cetuximab/ methotrexate
Drug: Methotrexate Injection — Administered intravenously
  Arms: cetuximab/ methotrexate

SUMMARY:
The objective of this study is to compare the efficacy and safety of MRG003 versus cetuximab/methotrexate as second/third line of therapy in patients with RM-SCCHN who have previously failed PD-1 (L1) inhibitors and platinum-based therapy.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter Phase III study to compare the efficacy and safety of MRG003 versus cetuximab/methotrexate as second/third line of therapy in patients with RM-SCCHN who have previously failed PD-1 (L1) inhibitors and platinum-based therapy. Approximately 180 patients will be enrolled, randomized, and stratified according to the following: Eastern Cooperative Oncology Group Performance Status (ECOG PS, 0 vs 1) and prior treatment with anti-EGFR mAb (yes vs no). For patients in the control group, cetuximab will be selected as comparator if no prior treatment with anti-EGFR mAb; otherwise, methotrexate will be selected.

After signing the informed consent and screened per inclusion/exclusion criteria, eligible patients will be randomized at a ratio of 1 : 1 and treated with MRG003 (2.3 mg/kg, IV, d1, Q3W) or cetuximab (400 mg/m2 for the first week and 250 mg/m2 for subsequent weeks, QW) / methotrexate (40 mg/m2, IV, QW) until disease progression, death, intolerable toxicity, withdrawal of consent, initiation of a new anti-tumor therapy, or other reasons leading to treatment discontinuation as specified by protocol.

ELIGIBILITY:
Inclusion Criteria:

- 1. Understands and provides written informed consent and willing to follow the requirements specified in protocol.

2. Age: ≥18 years and ≤75 years. 3. Life expectancy: ≥3 months. 4. Must have histologically or cytologically confirmed recurrent or metastatic squamous cell carcinoma of the head and neck (including oral cavity, oropharynx, hypopharynx, larynx) who had previously failed PD-1 (L1) inhibitors and platinum-based therapy (in combination or sequential). Prior therapies should be no more than 2 lines.

Note: If disease progression occurred during neoadjuvant/adjuvant treatment or concurrent radiotherapy, or within 6 months after treatment discontinuation, the anti-tumor therapies (including platinum-based chemotherapy, anti-EGFR monoclonal antibody, PD-1 (L1) inhibitors, etc.) during neoadjuvant/adjuvant treatment or concurrent radiotherapy is counted as one line of prior treatment. Discontinuation or dose reduction of one drug, or change of platinum- or fluorouracil-based agents or PD-1 (L1) inhibitors without disease progression is considered as the same line of treatment.

5. Must have at least one measurable lesion per RECIST v1.1. Previously irradiated lesion cannot be considered as target unless there is documented progression three months after the last treatment of radiotherapy.

6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 1) with no deterioration within 2 weeks prior to enrollment.

7. Adequate bone marrow function, defined as meeting all of the following criteria and having no transfusion therapy within 3 weeks (21 days) or growth factors (G-CSF, EPO, etc.) support within 2 weeks (14 days) prior to dosing:

• Hemoglobin (Hb) ≥ 9.0 g/dL (90 g/L)

• Absolute neutrophil count (ANC) ≥ 1,500/mcL (1.5 × 109/L)

• Total platelet count (PLT) ≥ 100,000/mcL (100 × 109/L) 8. Adequate hepatic function, defined as all of the following:

• Total bilirubin (TBIL) ≤ 1.5×ULN;

• Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN if no liver metastasis; ALT or AST ≤ 3.0×ULN in the presence of liver metastasis;

• Alkaline phosphatase (ALP) ≤ 1.5×ULN; ≤ 2×ULN in the presence of liver metastasis;

• Serum albumin ≥ 30 g/L 9. Coagulation: International Normalized Ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (APTT) ≤ 1.5×ULN (unless patient is receiving anticoagulant therapy whose anticoagulant level should be within the therapeutic range). The laboratory parameters should be closely monitored by investigator if the patient is on anticoagulation therapy.

10. Adequate renal function, defined as Creatinine ≤ 1.5×ULN or creatinine clearance rate (Ccr) ≥ 50 mL/min if Creatinine > 1.5×ULN (Creatinine clearance is calculated using the modified Cockcroft-Gault equation. Creatinine clearance can be calculated as Ccr = [(140-age) × body weight (kg) × (0.85 for women only)]/(72 × serum creatinine) if no local guidelines are available (without significant electrolyte imbalance that is not easily corrected).

11. Baseline Left Ventricular Ejection Fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO).

12. A negative serum or urine pregnancy test within 7 days prior to the first dose of study treatment (females of childbearing potential). If urine pregnancy test is positive or cannot be confirmed as negative, a confirmatory serum pregnancy test is required.

13. Patients, both females and males, of reproductive potential must agree to use adequate contraception during study treatment and for 180 days after the last treatment.

1. Females of childbearing potential (who are not surgically sterile or postmenopausal for < 1 year) who are willing to use adequate and reliable contraception such as avoidance of heterosexual activity, sterilization, oral contraceptives, injectable contraceptives, intrauterine devices, condoms, etc., during the study until 180 days after the last dose of study drug.
2. Male patients who are willing to use latex condoms during any sexual contact with females of childbearing potential during treatment until 180 days after the last treatment, even if vasectomy has been successfully performed. Reservation of semen specimen prior to the first dose of study treatment is recommended for fertile males for potential future conception.

   Exclusion Criteria:
   * 1. Grade ≥2 peripheral neuropathy per CTCAE v5.0. 2. Is expected to require surgery or any other form of systemic or local anti-tumor therapy during the study, including maintenance therapy or radiotherapy (including palliative therapy, except for palliative therapy for non-target lesions) for SCCHN.

     3. Received systemic chemotherapy within 3 weeks, small molecule targeted therapy within 2 weeks or 5 half-lives (whichever is longer), biological anti-tumor therapy, macromolecule targeted therapy or immunotherapy within 4 weeks before the first dose of study treatment, or major surgery (except for minor surgery within 2 weeks and fully recovered); radiotherapy (except radiotherapy for CNS, wash-out period ≥ 28 days is required) within 14 days before the first dose of study treatment.

     4. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with brain metastases may participate provided they are treated and stable, and do not have the following:
     * Progressive or new neurological deficits, seizures, evidence of increased intracranial pressure, vomiting, or headache;
     * Evidence of enlarging brain metastases by MRI at least 4 weeks prior to the first dose and corticosteroids is required for at least 14 days prior to study drug treatment.

       5. Residual toxicities (except alopecia, fatigue, and Grade 2 hypothyroidism) due to prior anti-tumor therapy (including immunotherapy, targeted therapy, chemotherapy or radiotherapy) or ≥ Grade 1 (CTCAE v5.0) clinically significant laboratory abnormality.

       6. Uncontrolled or poorly controlled cardiac dysfunction, including congestive heart failure (CHF) ≥ Grade 2 (CTCAE v5.0 or New York Heart Association classification), history of myocardial infarction, unstable angina pectoris, ventricular tachycardia or torsades de pointes, or cardiac rhythm loss requiring treatment within 6 months prior to enrollment, for example, QTcF > 450 ms in men, QTcF > 470 ms in women, in presence of complete left bundle branch block or third-degree atrioventricular block. QTcF = QT/ (RR^0.33).

       7. Pulmonary embolism or deep venous thrombosis (except for thrombosis caused by infusion port or PICC line) within 3 months prior to the first dose of study drug.

       8. Known history of malignancy (except for patients with cutaneous basal cell carcinoma, superficial bladder carcinoma, cutaneous squamous cell carcinoma, carcinoma in situ, or papillary thyroid carcinoma who have undergone curative surgery) unless the patient has received potentially curative therapy and has not had disease recurrence within 5 years prior to study treatment.

   Note: The 5-year recurrence-free time requirement does not apply to SCCHN patients enrolled in this study.

   9. Any serious or uncontrolled systemic disease, including uncontrolled or poorly controlled hypertension (e.g., systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg), diabetes mellitus (glycosylated hemoglobin (HbA1c) > 8%), etc.

   10. Patients with active bleeding, history of coagulopathy, or receiving coumarin anticoagulant therapy.

   11. Known allergic reactions to any component or excipients of MRG003 (citric acid monohydrate, sodium citrate dihydrate, trehalose dihydrate, sodium chloride, and polysorbate 80) or known allergic reactions to other anti-EGFR agents (including investigational drug) or to other monoclonal antibodies ≥ Grade 3.

   12. Known active hepatitis B or C. Active hepatitis B is defined as known positive HBsAg result and HBV DNA ≥ 500 IU/mL. Active hepatitis C is defined as known positive hepatitis C antibody result and known quantitative hepatitis C virus (HCV) RNA results greater than the lower limit of detection. Presence of other serious liver diseases, including chronic autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis, alcoholic liver disease, or nonalcoholic steatohepatitis (NASH).

   13. Concurrent, serious, uncontrolled infection or known infection with human immunodeficiency virus (HIV) (HIV antibody positive), or diagnosis of acquired immunodeficiency syndrome (AIDS); or uncontrolled autoimmune disease; or previous allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or previous solid organ transplantation.

   14. Active bacterial, viral, fungal, rickettsial, or parasitic infection requiring systemic anti-infection therapy (unless treated and resolved prior to study treatment).

   15. Received live-virus vaccines within 30 days prior to the first dose of study treatment. Seasonal influenza vaccines or approved COVID-19 vaccines that do not contain live virus are permitted if vaccinated more than 1 week before the first dose of study treatment.

   16. History of interstitial pneumonia, severe chronic obstructive pulmonary disease with respiratory failure, severe pulmonary insufficiency, symptomatic bronchospasm, etc.

   17. Patients who are receiving an immunologically based treatment for any reason, including chronic use of systemic steroids equivalent to > 10 mg/day of prednisone within 7 days prior to the first dose of study treatment or at any time during the study. Note: Use of inhaled or topical steroids or systemic corticosteroids equivalent to ≤ 10 mg/day prednisone is permitted, as is short-term use of corticosteroids at doses equivalent to > 10 mg/day prednisone (e.g., pre-medication prior to contrast).

   18. Uncontrolled pleural, abdominal, pelvic effusion or pericardial effusion that requires ≥ 1 drainage per month.

   19. Any patient with a positive pregnancy or is breast-feeding. Female and male patients who are not expected to use adequate contraception during treatment and for 180 days after the last dose of treatment.

   20. Any other disease or clinically significant abnormality in laboratory parameters, or serious medical or psychiatric illnesses/conditions, substance abuse disorder including alcoholism, which in the judgment of the Investigator might compromise the safety of the patient, integrity of the study, interfere with the patient participation in the study, or confound or compromise the study objectives and their interpretability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline to study completion (up to 24 months)
  OS is defined as the duration from the start of treatment to death of any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Baseline to study completion (up to 24 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Objective Response Rate (ORR) | Baseline to study completion (up to 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline to study completion (up to 24 months)
  DCR is defined as the proportion of subjects achieving CR, PR, and SD after treatment.
Duration of Response (DOR) | Baseline to study completion (up to 24 months)
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Treatment Related Adverse Events (TRAE) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial is considered related to the study drug.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Serious Adverse Events (SAEs) | Baseline to 90 days after the last dose of study treatment
  Adverse events that are difficult to deal with in clinical drug research
Quality of Life (QOL) scores | Baseline to study completion (up to 24 months)
  Quality of Life is a concept of comprehensive evaluation of the advantages and disadvantages of life. It mainly refers to the assessment of individual physiological, psychological and social functions, which is an important indicator of the effectiveness of medical and health care services.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, PhD, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No